CLINICAL TRIAL: NCT04169854
Title: Pre-emptive Topical Lidocaine 5% Plaster for Prevention of Post-craniotomy Pain : a Protocol for a Randomized, Triple Blind, Placebo-controlled Trail
Brief Title: Pre-emptive Topical Lidocaine 5% Plaster for Prevention of Post-craniotomy Pain
Acronym: EASY
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Clinical Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY 2019-122-02
Record Dates: First submitted 2019-11-11; First posted 2019-11-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Postoperative Pain; Lidocaine
Keywords: Postoperative Pain; Postcraniotomy Pain; Lidocaine Patch
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine; Transdermal Patch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine Patch (Experimental): Surgeons will be asked to mark the planned incisions site 3 days before craniotomy. The masked Lidocaine 5% patch will be applied to cover the insicion mark as well as the head-holders sites within 6:00 P.M. to 6:00 A.M. for 3 consecutive preoperative days.
  Interventions: Drug: Lidocaine 5% patch
- Placebo (Placebo Comparator): Surgeons will be asked to mark the planned incisions site 3 days before craniotomy. The masked placebo patch will be applied to cover the insicion mark as well as the head-holders sites within 6:00 P.M. to 6:00 A.M. for 3 consecutive preoperative days.
  Interventions: Drug: Placebo patch

INTERVENTIONS:
Drug: Lidocaine 5% patch — The Lidocaine 5% Patch will be applied to cover the marked incision site and head-holders sites for 3 consecutive preoperative days between 6:00 P.M. to 6:00 A.M.. Research assistants will be responsible for instructing patients to cover the patches correctly.
  Arms: Lidocaine Patch
Drug: Placebo patch — The Placebo Patch will be applied to cover the marked incision site and head-holders sites for 3 consecutive preoperative days between 6:00 P.M. to 6:00 A.M.. Research assistants will be responsible for instructing patients to cover the patches correctly.
  Arms: Placebo

SUMMARY:
Postcraniotomy pain remains a common phenomenon in the neurosurgery field. Managements for postcraniotomy pain are to be standardised and optimized. In the proposed study, the investigators aim to provide a novel regional non-invasive prophylactic strategy for postcraniotomy pain by utilizing Lidocaine 5% plaster.

DETAILED DESCRIPTION:
Postcraniotomy pain remains a common phenomenon in the neurosurgery field. Insufficient control of postcraniotomy pain may lead to unexpected clinical outcomes. The current management for postcraniotomy pain mainly involves systemic intravenous or oral medication and regional anaesthetic injection.

The investigators intend to compare pre-emptive lidocaine 5% plaster incision covering to a placebo for prophylaxis of postcraniotomy pain. In the proposed study, the effectiveness and safety of lidocaine 5% plaster for postcraniotomy pain control will be examined compared with those of placebo. The investigators aim to provide a novel regional non-invasive prophylactic strategy for postcraniotomy pain.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 or older
* American Society of Anesthesiologists status I or II
* Registered for elective craniotomy
* Informed consent for participation in the trial

Exclusion Criteria:

* Allergy to lidocaine or the hydrogel plaster
* Chronic headache, craniofacial pain or neuralgia
* Glasgow Coma Scale less than 15
* Current or previous cardiovascular or cerebrovascular accident
* Expected delayed recovery or extubation
* Uncontrolled arrhythmia
* History of intracranial operation
* Emergency or revision craniotomy
* Mental illness, psychiatric drug use or alcohol abuse
* Failure to understand the use of a 100 mm VAS or the PCA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 24 hours after craniotomy
  Pain intensity will be examined using the 0 - 100 mm visual analogue scale scores, where '0' represents 'no pain' ,and '100' represents 'the most severe pain'.

SECONDARY OUTCOMES:
Pain intensity | 1, 4, 6, 12, 48 and 72 hours after craniotomy
  Pain intensity will be examined using the 0 - 100 mm visual analogue scale scores, where '0' represents 'no pain' ,and '100' represents 'the most severe pain'.
Time interval to analgesics | 0-72 hours after craniotomy
  Time interval from the end of craniotomy to the first press of the PCA device and to the first rescue analgesic administration
Cumulative butorphanol | 24, 48 and 72 hours after craniotomy
  he cumulative butorphanol consumption through the PCA device
Cumulative intraoperative analgesics consumption | During the craniotomy
  Cumulative intraoperative opioids consumption
Length of hospital stay | within 3 months
  Time length from admission to leaving the hospital
Lidocaine 5% plaster safety (local) | 3 preoperative days
  Rate of patients with local adverse event as graded using NCI-CTCAE V4.0
Lidocaine 5% plaster safety (systemic) | 3 preoperative days
  Rate of patients with systemic adverse event as graded using NCI-CTCAE V4.0
Pittsburgh Sleep Quality Index (PSQI) | first 3 days after craniotomy.
  The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions which measures seven aspects of sleep: (1) subjective sleep quality, (2) sleep latency, (3) sleep duration, (4) habitual sleep efficiency, (5) sleep disturbances, (6) use of sleeping medication, and (7) daytime dysfunction. The 19 self-rated items are combined to form seven component scores, each of which has a range of 0-3 points (0 indicates no difficulty, while 3 indicates severe difficulty). The seven component scores are then summed to yield one global score, with a range of 0-21 points (0 indicating no difficulty, and 21 indicating severe difficulties in all the seven areas of sleep quality).

CONTACTS AND LOCATIONS:
Overall Officials: Fang Luo, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gottschalk A, Berkow LC, Stevens RD, Mirski M, Thompson RE, White ED, Weingart JD, Long DM, Yaster M. Prospective evaluation of pain and analgesic use following major elective intracranial surgery. J Neurosurg. 2007 Feb;106(2):210-6. doi: 10.3171/jns.2007.106.2.210. PMID 17410701
- [Background] Mordhorst C, Latz B, Kerz T, Wisser G, Schmidt A, Schneider A, Jahn-Eimermacher A, Werner C, Engelhard K. Prospective assessment of postoperative pain after craniotomy. J Neurosurg Anesthesiol. 2010 Jul;22(3):202-6. doi: 10.1097/ANA.0b013e3181df0600. PMID 20479664
- [Background] Artime CA, Aijazi H, Zhang H, Syed T, Cai C, Gumbert SD, Ferrario L, Normand KC, Williams GW, Hagberg CA. Scheduled Intravenous Acetaminophen Improves Patient Satisfaction With Postcraniotomy Pain Management: A Prospective, Randomized, Placebo-controlled, Double-blind Study. J Neurosurg Anesthesiol. 2018 Jul;30(3):231-236. doi: 10.1097/ANA.0000000000000461. PMID 29117012
- [Background] Licina A, Russell J, Silvers A, Jin X, Denny J. Subcutaneous sumatriptan for the treatment of postcraniotomy pain (SUPS trial): protocol for a randomised double-blinded placebo controlled trial. BMJ Open. 2019 Aug 18;9(8):e032388. doi: 10.1136/bmjopen-2019-032388. PMID 31427345
- [Background] Hassani E, Mahoori A, Sane S, Tolumehr A. Comparison the effects of paracetamol with sufentanil infusion on postoperative pain control after craniotomy in patients with brain tumor. Adv Biomed Res. 2015 Mar 4;4:64. doi: 10.4103/2277-9175.152610. eCollection 2015. PMID 25821764
- [Derived] Han X, Yang Y, Ren T, Ji N, Luo F. Efficacy of Preemptive Topical Lidocaine 5% Plaster in the Prevention of Post-Craniotomy Pain, a Randomized Clinical Trial. J Pain Res. 2024 Dec 13;17:4251-4261. doi: 10.2147/JPR.S499264. eCollection 2024. PMID 39691748